CLINICAL TRIAL: NCT00709020
Title: A Translational Breast Cancer Prevention Trial of Mushroom Powder in Postmenopausal Breast Cancer Survivors
Brief Title: White Button Mushroom Extract in Preventing the Recurrence of Breast Cancer in Postmenopausal Breast Cancer Survivors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07213; P30CA033572 (NIH); CHNMC-07213; CDR0000599204 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Cancer Survivor
Keywords: cancer survivor; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Flow Cytometry; Chromatography, High Pressure Liquid; Mass Spectrometry; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- White Button Mushroom Extract (Experimental)
  Interventions: Drug: white button mushroom extract; Other: flow cytometry; Other: high performance liquid chromatography; Other: laboratory biomarker analysis; Other: mass spectrometry; Other: pharmacogenomic studies; Other: pharmacological study

INTERVENTIONS:
Drug: white button mushroom extract — Dose escalation with six evaluable subjects per dose level. Doses begin at 5 g/day, then 8 g/day, then 10 g/day then 13 g/day.
Other: flow cytometry — Performed on blood samples taken day -14 and -7 prior to treatment and days 1, 8, 15, 29, 57 and 85 of treatment.
Other: high performance liquid chromatography — Performed on blood samples taken day -14 and -7 prior to treatment and days 1, 8, 15, 29, 57 and 85 of treatment.
Other: laboratory biomarker analysis — Performed on blood samples taken pre-treatment on day 1 and on day 85 after treatment.
Other: mass spectrometry — Performed on blood samples taken day -14 and -7 prior to treatment and days 1, 8, 15, 29, 57 and 85 of treatment.
Other: pharmacogenomic studies — Performed on blood samples taken on days 1, 8, 15, 29, 57 and 85 of treatment.
Other: pharmacological study — Performed on blood samples taken pre-dose and at 0.25, 0.5, 0.75, 1, 2, 4 and 6 hours after White Button Mushroon extract on day 1 of treatment and pre-dose on days 8, 15, 29, 57 and 85 after start of treatment.

SUMMARY:
RATIONALE: White button mushroom extract may stop or delay the recurrence of breast cancer in postmenopausal breast cancer survivors.

PURPOSE: This phase I trial is studying the side effects and best dose of white button mushroom extract in preventing the recurrence of breast cancer in postmenopausal women who are breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To show that a whole food extract of white button mushrooms (WBM) can inhibit aromatase-induced estrogen biosynthesis in postmenopausal women who are breast cancer survivors (BCS).
* To determine the optimal daily dose of WBM needed to induce aromatase inhibition of estrogen biosynthesis in these patients.
* To determine the bioavailability of C-18 unsaturated fatty acids, which are thought to moderate the anticancer effects of WBM.

Secondary

* To determine the safety and tolerability of WBM in humans via serial comprehensive symptom questionnaires, pre- and post-treatment markers of bone metabolism, and pre- and post-treatment comprehensive lipid panels.
* To explore potential alternate antitumor mechanisms, specifically the effect of WBM on cytokines as well as innate and adaptive cellular immunity.
* To describe barriers experienced in recruitment of ethnically diverse subjects from the community into a secondary prevention BCS trial utilizing a dietary supplement intervention in an effort to enhance feasibility of a subsequent phase II trial.

OUTLINE: This is a dose-escalation study.

Patients receive oral white button mushroom extract twice daily for 12 weeks in the absence of a second primary ductal carcinoma in situ, invasive breast cancer, or unacceptable toxicity.

Patients undergo blood and urine sample collection at baseline and periodically during treatment for pharmacokinetic, pharmacodynamic, and immunologic correlative studies. Blood and urine samples are analyzed for concentrations of C-18 unsaturated fatty acids (CUFA) by high-performance liquid chromatography tandem-mass spectrometry. Blood samples are also analyzed for anti-aromatase activity by ex vivo plasma aromatase inhibition assays; circulating sex steroid hormones by radioimmunoassay; serum immune cytokine levels by multiplex cytokine analyses; immunophenotyping, NK-cell activation status, and NK-cell function by multiparameter flow cytometry; lipid levels by lipid assays; and biochemical markers of bone metabolism by bone metabolism marker assays. DNA, RNA, and plasma samples are stored for post-trial pharmacogenomic studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Prior diagnosis of infiltrating carcinoma of the breast ≥ 5 years prior to study entry
  * Prior diagnosis of ductal carcinoma in situ
* No evidence of disease
* Completed all cancer therapy, with the exception of reconstructive surgery, at least 6 months prior to study entry
* Meets one of the following criteria:

  * Normal mammogram within 1 year of study entry
  * Underwent bilateral mastectomy and has been in remission for 5 years, as documented by an oncologist
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,500/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Postmenopausal, defined as any of the following:

  * Continuous absence of menstruation for 12+ months
  * Status post bilateral oophorectomy
  * Status post hysterectomy with follicle-stimulating hormone in menopausal range
* Creatinine ≤ 1.5 times upper limit of normal (ULN) or less
* Total bilirubin ≤ 1.5 times ULN
* AST and ALT < 2 times ULN
* No allergy to mushrooms
* No personal history of any invasive cancer, other than breast cancer, or squamous cell or basal cell skin cancer
* No osteoporosis, defined as a bone-mineral density T-score of < -2.5 on dual-energy x-ray absorptiometry scan
* No major systemic infections or other major medical illnesses of the cardiovascular, respiratory, or digestive system

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 months since prior and no concurrent hormone-modifying medications, including any of the following:

  * Oral contraceptives
  * Hormone replacement
  * Selective estrogen receptor modifiers
  * Other aromatase inhibitors
  * Gonadotropic-releasing hormone modifiers
* At least 1 month since prior and no other concurrent mushroom extracts or DHEA as a dietary supplement
* No concurrent therapy, except continued medications for unrelated illness that are not excluded, and necessary medications for unrelated acute illnesses that may occur during the study (e.g., cold, flu, or infection)
* No more than 3 concurrent servings per week of the following foods:

  * Flaxseeds and flaxseed meal
  * High-energy bars or diet bars containing soy or soy protein
  * Liquid-nutrition drinks containing soy or soy protein (e.g., Odwalla Future Shake or Ensure Plus)
  * Miso soup
  * Natto
  * Packaged mixed dishes with soy or tofu (e.g., lasagna, burritos, or stir-fry)
  * Cooked soybeans or edamame (i.e., green soybeans)
  * Roasted soy nuts
  * Soymilk, regular or low-fat, plain or flavored
  * Soy cheese, such as cheddar, mozzarella, cram cheese, or parmesan (includes all foods made with soy cheese)
  * Soy protein powders (e.g., performance or body-builder powders)
  * Soy yogurt, all types
  * Soy sauce, tamari, teriyaki sauce, Szechuan sauce, or hoisin sauce
  * Soy ice cream, tofutti, or other soy desserts
  * Tempeh, all types
  * Tofu, all types, including low-fat, flavored, marinated, and smoked
  * Tofu or soy breakfast sausage, bacon, or other breakfast meat
  * Tofu or soy cold cuts, hot dogs, or other deli meat substitutes
  * Veggie soy or tofu burger, ground meat substitute (texturized vegetable protein), or soy or tofu, chicken, or turkey
* Concurrent supplemental calcium and/or vitamin D and bisphosphonates allowed provided doses remain constant throughout the run-in and treatment portions of the trial

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of white button mushroom extract (WBM) in reducing serum estradiol (E2) | Baseline prior to treatment, days 8, 15, 29, 57 and 85 after the start of treatment.
Serum sex steroid hormone levels | Baseline prior to treatment, days 8, 15, 29, 57 and 85 after the start of treatment.
Optimal daily dose of WBM | 1 year after completion of the study
Pharmacokinetics of C-18 unsaturated fatty acids (CUFA) as measured by high-performance liquid chromatography tandem-mass spectrometry | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 4 and 6 hours after White Button Mushroon extract on day 1 of treatment and pre-dose on days 8, 15, 29, 57 and 85 after start of treatment.
Pharmacodynamics of WBM as measured by ex vivo plasma aromatase inhibition assays | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 4 and 6 hours after White Button Mushroon extract on day 1 of treatment and pre-dose on days 8, 15, 29, 57 and 85 after start of treatment.

SECONDARY OUTCOMES:
Safety and tolerability of WBM as assessed by NCI CTCAE v3.0, symptom logs, bone metabolism markers, and pre- and post-treatment comprehensive lipid panels | 4 months after completion of treatment
Effect of WBM on cytokines as measured by multiplex cytokine analyses | Day -14 and Day -7 before first treatment, Day 1, 8, 15, 29, 57 and 85 after treatment begins.
Effect of WBM on innate and adaptive cellular immunity as measured by immunologic assays | Day -14 and Day -7 before first treatment, Day 1, 8, 15, 29, 57 and 85 after treatment begins.
Barriers to recruitment of ethnically diverse patients from the community | 4 months after completion of treatment
Dietary sources of CUFA as measured by food frequency questionnaires | Day -14 before treatment begins, day 1, 29, 57 and 85 after treatment begins
Bone metabolism markers (i.e., serum procollagen type-1 propeptide and urine N-telopeptide crosslinks) | Day 1 of treatment and day 85 of treatment
Fasting lipids (i.e., total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides) | Day 1 of treatment and day 85 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shiuan Chen, PhD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California